CLINICAL TRIAL: NCT06250374
Title: Assessment of the Cerebral Perfusion During the Period of Deep Hypothermia at 18°C in Patient Undergoing Pulmonary Endarterectomy Surgery.
Acronym: HYPO-TEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A00270-45
Record Dates: First submitted 2024-01-12; First posted 2024-02-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hypothermia; Cerebral Perfusion; Transcranial Doppler Ultrasound; Pulmonary Hypertension
Keywords: Pulmonary endarterectomy; cerebral perfusion; Hypothermia; Transcranial doppler ultrasound; Cardiopulmonary bypass
MeSH Terms: conditions — Hypothermia; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with thromboendarterectomy surgery (Experimental): Anesthesia was induced with sufentanil 0.3 g/kg, etomidate 0.3-0.4 mg/kg, rocuronium 0.4 mg/kg and maintained with continuous infusion Propofol and sufentanil. A pulmonary arterial catheter was inserted in all patients. Patients were cooled by means of the oxygenator heat exchanger at a rate of one degree Celsius every three minutes. Rewarming was achieved at a rate of one degree Celsius every five to ten minutes.
  The following measures were performed:
  Measure 1: In normo-thermia after induction of general anesthesia Measure 2: On CPB, before circulatory arrest and in hypothermia at 18-20°C Measure 3: On bypass, after circulatory arrest and in hypothermia at 18-20°C Measure 4: At the end of the procedure, after weaning from the bypass and in normothermia.
  For each measure mean arterial pressure, cardiac output, PaCO2, pH, bilateral NIRS value were also recorded.
  Interventions: Procedure: Bilateral trans-cranial Doppler ultrasound

INTERVENTIONS:
Procedure: Bilateral trans-cranial Doppler ultrasound — Velocity measurements in the middle cerebral artery are made using an ultrasound probe applied to the patient's temple during surgery.

SUMMARY:
Cardiopulmonary bypass (CPB) surgery present risk of acute postoperative neurological complications. These complications are most often postoperative cognitive dysfunction (confusion, cognitive disorders, executive disorders) with a prevalence of up to 40% at 5 years, and ischemic (stroke) with an incidence of between 0.4 and 14%. The causes are usually multifactorial, but altered cerebral perfusion during CPB surgery is an important prognostic factor. Data regarding the effect of deep hypothermia on cerebral perfusion during CPB in adult are scarce. Currently, aortic arch replacement following aortic dissection or aneurysm, and pulmonary artery endarterectomy (PAE) in the treatment of pulmonary hypertension of post embolic origin are performed under deep hypothermia.

In this latter indication, the need to obtain a completely bloodless operating field necessitates complete circulatory arrest during short period of time to enable the surgeon to optimally remove the clot materials located into the pulmonary arteries.

To protect the brain and avoid irreversible brain injury during circulatory arrest(s), body temperature is lowered at 18-20°C. Deep hypothermia can lead to significant arterial vasoconstriction, which can reduce the blood supply to the brai. It also increases the solubility of CO2 in the blood, leading to respiratory alkalosis, which can also lead to vasoconstriction of cerebral vessels, increasing the risk of ischemic lesions.

In adult there is no consistent data on the cerebral perfusion during PAE surgery under deep hypothermia at 18-20°C. Animal studies showed that cerebral regulation seems to be preserved under these conditions. A better understanding of the effect of deep hypothermia on cerebral perfusion during PAE surgery is essential to adapt our management to limit the occurrence of postoperative neurological complications.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for pulmonary artery thromboendarterectomy surgery.
* Patient with free, written and informed consent.
* Patient affiliated to a social security scheme (beneficiary or beneficiary's beneficiary).
* French-speaking patient.

Exclusion Criteria:

* Patient refusing to participate in the study.
* Patient under guardianship.
* Patient deprived of liberty.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
Assessment of cerebral blood perfusion during deep hypothermia | M1: Baseline-normothermia after induction of general anesthesia (H0) M2: During CPB-at 18°C-before cardiac arrest (H2) M3: After cardiac arrest-at 18°C before (H4) M4: End of surgery-normothermia (H6)
  Cerebral blood perfusion during deep hypothermia (18-20°C) will be assessed by measuring mean blood flow velocities in the middle cerebral arteries (MCAs) using trans-cranial Doppler ultrasound (DTC) at different time of the surgery (Four measures in total). All measure are performed during the time of the surgery. The first measure (M1) is baseline to which the other measure will be compared to.

SECONDARY OUTCOMES:
Correlation between NIRS and middle cerebral arteries velocity values for each measure. | M1: Baseline-normothermia after induction of general anesthesia (H0) M2: During CPB-at 18°C-before cardiac arrest (H2) M3: After cardiac arrest-at 18°C before (H4) M4: End of surgery-normothermia (H6)
  For each measure of middle cerebral arteries blood flow velocity performed during the surgery, the value of the near infrared spectroscopy (NIRS) is recorded. A total of four measures is performed during the time of the surgery.
Seek for post-circulatory arrest hyperemia | M2: During CPB after cooling at 18°C before cardiac arrest (H2). M3: After cardiac arrest at 18°C before rewarming period (H4).
  Comparison of the middle cerebral arteries blood flow velocities during the period of hypothermia, before and after cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Marie Lannelongue, Le Plessis-Robinson, France

REFERENCES:
- [Background] Liu Y, Chen K, Mei W. Neurological complications after cardiac surgery: anesthetic considerations based on outcome evidence. Curr Opin Anaesthesiol. 2019 Oct;32(5):563-567. doi: 10.1097/ACO.0000000000000755. PMID 31145196
- [Background] Brown CH 4th, Neufeld KJ, Tian J, Probert J, LaFlam A, Max L, Hori D, Nomura Y, Mandal K, Brady K, Hogue CW; Cerebral Autoregulation Study Group; Shah A, Zehr K, Cameron D, Conte J, Bienvenu OJ, Gottesman R, Yamaguchi A, Kraut M. Effect of Targeting Mean Arterial Pressure During Cardiopulmonary Bypass by Monitoring Cerebral Autoregulation on Postsurgical Delirium Among Older Patients: A Nested Randomized Clinical Trial. JAMA Surg. 2019 Sep 1;154(9):819-826. doi: 10.1001/jamasurg.2019.1163. PMID 31116358